CLINICAL TRIAL: NCT00042653
Title: A Placebo-controlled, Double-blind, Multicenter Study to Assess the Efficacy and Safety of an Oral Calcimimetic Agent (AMG 073) in Secondary Hyperparathyroidism of Chronic Kidney Disease (Hemodialysis and Peritoneal Dialysis)
Brief Title: A Study of an Investigational Medication for the Treatment of Secondary Hyperparathyroidism in Patients on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20000188
Record Dates: First submitted 2002-08-02; First posted 2002-08-06 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Secondary Hyperparathyroidism; End Stage Renal Disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AMG 073 (Experimental): AMG 073
  Interventions: Drug: AMG 073
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 30 mg of placebo taken once daily orally 60 mg of placebo taken once daily orally 90 mg of placebo taken once daily orally 120 mg of placebo taken once daily orally 180 mg of placebo taken once daily orally
  Arms: Placebo
Drug: AMG 073 — 30 mg of AMG 073 taken once daily orally 60 mg of AMG 073 taken once daily orally 90 mg of AMG 073 taken once daily orally 120 mg of AMG 073 taken once daily orally 180 mg of AMG 073 taken once daily orally
  Arms: AMG 073

SUMMARY:
This 6 month study will assess an investigational medication for patients on dialysis with secondary hyperparathyroidism. The study will look at the effects on parathyroid hormone, calcium and phosphorus levels.

ELIGIBILITY:
Patients must be receiving hemodialysis; have elevated parathyroid hormone levels; not be pregnant or nursing; and not have had a heart attack in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2002-05; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of AMG 073 compared with placebo by determining the proportion of subjects with a mean intact parathyroid hormone (iPTH) value <= 250 pg/mL (26.5 pmol/L) during the efficacy assessment phase. | Efficacy Assessment phase - final 10 weeks of study

SECONDARY OUTCOMES:
To evaluate the efficacy of AMG 073 compared with placebo by determining: the proportion of subjects with a reduction from baseline in mean iPTH of >= 30% during the efficacy assessment phase | Efficacy Assessment phase - final 10 weeks of study
To evaluate the efficacy of AMG 073 compared with placebo by determining: percentage change from baseline in iPTH during the efficacy assessment phase | Efficacy Assessment phase - final 10 weeks of study
To evaluate the safety of AMG 073 compared with placebo | Entire study - 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Lindberg JS, Culleton B, Wong G, Borah MF, Clark RV, Shapiro WB, Roger SD, Husserl FE, Klassen PS, Guo MD, Albizem MB, Coburn JW. Cinacalcet HCl, an oral calcimimetic agent for the treatment of secondary hyperparathyroidism in hemodialysis and peritoneal dialysis: a randomized, double-blind, multicenter study. J Am Soc Nephrol. 2005 Mar;16(3):800-7. doi: 10.1681/ASN.2004060512. Epub 2005 Feb 2. PMID 15689407
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_38_AMG_073_20000188.pdf
- See also: FDA-approved Drug Labeling — http://www.sensipar.com/